CLINICAL TRIAL: NCT05814133
Title: Prospective Clinical Trial To Evaluate The Thulium Fiber Laser For The Ureteroscopic Treatment Of Nephrolithiasis
Brief Title: Thulium Fiber Laser Prospective Trial
Acronym: TFL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: University of British Columbia (Other); Columbia University (Other); University of California, San Diego (Other); Mayo Clinic (Other); Ohio State University (Other); Vanderbilt University (Other); The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-11370
Record Dates: First submitted 2023-03-09; First posted 2023-04-14 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Kidney Stone
Keywords: ureteroscopy; lithotripsy; thulium fiber laser
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lithotripsy (Experimental): Ureteroscopy with lithotripsy using the Thulium Fiber Laser
  Interventions: Device: Thulium Fiber Laser

INTERVENTIONS:
Device: Thulium Fiber Laser — Thulium Fiber Laser will be used to break renal stones < 2 cm into fragments small enough to remove or pass spontaneously through the ureter.

SUMMARY:
This is a multi-center, prospective clinical trial to assess the effect of TFL for the lithotripsy of kidney stones.

DETAILED DESCRIPTION:
Flexible ureteroscopy is considered the first-line therapy for renal stones < 2 cm. The Holmium: YAG laser (Ho:YAG) is established as gold standard in urology practice. Despite its limitations, it is widely used to break stones into fragments small enough to remove or pass spontaneously through the ureter. Advances in the understanding of laser energy delivery have led to the recent commercialization of the 'Thulium Fiber Laser' (TFL) with unique characteristics and promising improvements of ablation efficiency, dusting capacity, operating time and deflection. A a multi-center, prospective clinical trial to further assess those advantages for the lithotripsy of kidney stones will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Solitary renal stone 8 to 20 mm in size or in the case of multiple stones the conglomerate diameter of 8-20 mm is required
* Must be a suitable operative candidate for flexible ureteroscopy per urologic guidelines
* Must be 18 years or older
* Must be able to give consent
* Bilateral ureteroscopy will be permitted but only the first side will be included in the study

Exclusion Criteria:

* Concomitant stones in the ureter
* Prior ipsilateral upper urinary tract reconstructive procedures or history of ipsilateral ureteral stricture
* Prior radiotherapy to the abdomen or pelvis
* Neurogenic bladder or spinal cord injury
* Pregnancy
* Untreated Urinary Tract Infection (UTI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Mean total operative time | during the procedure
  Total operative time during the ureteroscopic treatment of renal stones using a laser dusting technique.

SECONDARY OUTCOMES:
Rate of stone retropulsion | during the procedure
  Review of the procedure video recording to assess stone retropulsion occurence during stone lithotripsy

OTHER OUTCOMES:
Mean length of hospitalization | From day and time of admission to day and time of discharge
  Length of hospitalization (in days) for the procedure will be recorded for each patient
Rate of postoperative complications | at 6 weeks
  Medical chart review will be done to assess the occurence of post-operative complications
Rate of stone free status | at 6 weeks
  Post-operative CT imaging will be reviewed to assess the occurence of ''stone free status''
Rate of need for ancillary procedures | at 6 weeks
  Medical chart review will be done to assess the occurence of an additional ureteroscopy need to treat patients
Mean perceived workload score | immediately after the procedure
  Effects of TFL technology on reducing surgeon perceived workload will be assessed by completing the National Aeronautics and Space Administration (NASA) Task Load Index. The tool allows to determine the subjective mental workload (MWL) of a participant while they are performing a task.The participants self-rate on a scale of 1 (low) to 20 (high). The higher the score, the worst is the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Naeem Bhojani, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Background] Kronenberg P, Traxer O. Update on lasers in urology 2014: current assessment on holmium:yttrium-aluminum-garnet (Ho:YAG) laser lithotripter settings and laser fibers. World J Urol. 2015 Apr;33(4):463-9. doi: 10.1007/s00345-014-1395-1. Epub 2014 Sep 4. PMID 25185524
- [Background] Nazif OA, Teichman JM, Glickman RD, Welch AJ. Review of laser fibers: a practical guide for urologists. J Endourol. 2004 Nov;18(9):818-29. doi: 10.1089/end.2004.18.818. PMID 15659912
- [Background] Khusid JA, Khargi R, Seiden B, Sadiq AS, Atallah WM, Gupta M. Thulium fiber laser utilization in urological surgery: A narrative review. Investig Clin Urol. 2021 Mar;62(2):136-147. doi: 10.4111/icu.20200467. PMID 33660440
- [Background] Kronenberg P, Hameed BZ, Somani B. Outcomes of thulium fibre laser for treatment of urinary tract stones: results of a systematic review. Curr Opin Urol. 2021 Mar 1;31(2):80-86. doi: 10.1097/MOU.0000000000000853. PMID 33470684
- [Background] Traxer O, Corrales M. Managing Urolithiasis with Thulium Fiber Laser: Updated Real-Life Results-A Systematic Review. J Clin Med. 2021 Jul 30;10(15):3390. doi: 10.3390/jcm10153390. PMID 34362169
- [Background] Law KE, Lowndes BR, Kelley SR, Blocker RC, Larson DW, Hallbeck MS, Nelson H. NASA-Task Load Index Differentiates Surgical Approach: Opportunities for Improvement in Colon and Rectal Surgery. Ann Surg. 2020 May;271(5):906-912. doi: 10.1097/SLA.0000000000003173. PMID 30614878
- See also: Chew * Ben H., Knudsen BE, Molina WR. Mp79-19 comparison of dusting and fragmenting using the new super pulse thulium fiber laser to a 120w holmium:yag laser. Journal of Urology. 2019 Apr;201(Supplement 4):e1159-60. — http://www.urotoday.com/conference-highlights/aua-2019-annual-meeting/aua-2019-stone-disease/112422-aua-2019-comparison-of-dusting-and-fragmenting-using-the-new-super-pulse-thulium-fiber-laser-to-a-120w-holmium-yag-laser.html